CLINICAL TRIAL: NCT02459925
Title: MOMS Partnership-Community-Based Hubs for Maternal Mental Health and Workforce Development, New Haven MOMS Partnership- CT Dept of Social Services Block Grant
Brief Title: MOMS Hubs- CT Dept of Social Services Block Grant
Acronym: MOMS-Hubs
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to funding that was never obtained, the MOMS Grow arm was not completed.
Sponsor: Yale University (Other)
Collaborators: Clifford Beers Clinic (Unknown); City of New Haven- Health Department (Unknown); New Paradigms Consulting (Unknown); National Diaper Bank Network (Unknown); The New Haven Diaper Bank (Unknown); Third Sector Capital Partners (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1409014610
Record Dates: First submitted 2015-04-08; First posted 2015-06-02 (Estimated); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT- Mental Health Program (Active Comparator): Cognitive Behavioral Therapy. Manualized Stress Management class; brief individual behavioral counseling.
  Interventions: Behavioral: CBT- Mental Health Program
- MOMS GROW (Active Comparator): MOMS GROW (Generating Real Opportunities for Work) Teaching, coaching, and supportive services for participants as they navigate their journeys to sustainable employment that pays a family-supporting wage.
  Interventions: Behavioral: MOMS GROW

INTERVENTIONS:
Behavioral: CBT- Mental Health Program — Manualized Stress Management class; brief individual behavioral counseling.
  Arms: CBT- Mental Health Program
Behavioral: MOMS GROW — MOMS GROW (Generating Real Opportunities for Work) Teaching, coaching, and supportive services for participants as they navigate their journeys to sustainable employment that pays a family-supporting wage.
  Arms: MOMS GROW

SUMMARY:
The MOMS Partnership aims to create "MOMS Zones" in New Haven neighborhoods where the hardest to reach families live. These "MOMS Zones" will have two unique features: (1) a MOMS "Hub" to deliver centralized mental health and family economic success services to the hardest to reach families living in New Haven's most impoverished neighborhoods, as measured by actual socio-economic status as well as by access to resources; (2) a neighborhood workforce of Community Mental Health Ambassadors (CMHAs--mothers who themselves live in New Haven). The MOMS Workforce Program and MOMS Mental Health Program will be offered at all three Hubs.

DETAILED DESCRIPTION:
The MOMs workforce program will involve teaching, coaching, and supportive services for participants as they navigate their journeys to sustainable employment that pays a family-supporting wage. Participants will be guided through an individualized progression of services designed to increase their employability, to increase their ability to earn higher incomes in career-track employment, and to improve their chances of retaining jobs and advancing in them.

The MOMS Mental Health program centers around a manualized Stress Management Course 8-class group treatment, delivered once per week. The course was adapted from "The Mother and Child Course" by Munoz and Le (2011) for the population of New Haven mothers who are served by the MOMS Partnership.

ELIGIBILITY:
Inclusion criteria are as follows:

* Participant is a woman raising a child or adolescent under 18 years of age. The child/adolescent may be her biological offspring or in her custody due to adoption or foster care. Care arrangements may be legally sanctioned or informal, as is common in New Haven families. Thus, the eligible participant may be a sister, aunt, grandmother, or other female responsible for the daily care of children.
* Participant currently resides within the city limits of New Haven, CT.
* Participant resided within County of New Haven, CT on October 29, 2012.
* Participant's income is at or below 325% of the Federal poverty income.
* Participant is a U.S. citizen.
* Participant's score on CES-D > 16.

Exclusion criteria are as follows:

* Signs or symptoms of active psychosis or active suicidality will be a basis for exclusion in the study.
* Lack of proficiency in English.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2015-04-22 (Actual); Primary Completion 2017-05-25 (Actual); Study Completion 2017-05-25 (Actual)

PRIMARY OUTCOMES:
Improvement in Center for Epidemiologic Studies Depression (CED-D) Scale | 6 months
  Reduced CES-D Score (CES-D score goal <16)
Improvement in work readiness skills | 6 months
  Reduced CASAS score

CONTACTS AND LOCATIONS:
Overall Officials: Megan V Smith, DrPH, Principal Investigator — Yale University
Locations (4):
- United States (4):
  - Boys & Girls Club of New Haven, New Haven, Connecticut
  - Center for Wellbeing of Women and Mothers, Dept. of Psychiatry, Yale University, New Haven, Connecticut
  - Stop & Shop, New Haven, Connecticut
  - West Rock Author's Academy, New Haven, Connecticut